CLINICAL TRIAL: NCT01265680
Title: Single High Dose Erythropoietin Obviates Transfusions: an Independent, Blinded, Prospective Randomized Study in Heart Surgery Population.
Brief Title: Blood Sparing Strategies: Single Shot High Dose Erythropoietin Two Days Before Heart Surgery
Acronym: SHOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Principal Investigator, Luca Weltert, Project Leader Luca Weltert, Cardiochirurgia E.H.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-05
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Blood Transfusion
Keywords: Blood Transfusion; Heart surgery; Erythropoietin; HRE
MeSH Terms: interventions — Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Experimental): 80.000 UI of Human Recombinant Erythropoietin and intravenous iron at time of arrival at the hospital
  Interventions: Drug: Erythropoietin
- Control (No Intervention): No added administration other than our standard of care.

INTERVENTIONS:
Drug: Erythropoietin — 80.000 UI of Human Recombinant Erythropoietin and intravenous iron at time of arrival at the hospital.
  Other Names: Eprex
  Arms: Erythropoietin

SUMMARY:
All patients operated on at the European Hospital Heart surgery Division will be randomized to either single dose 80.000 UI of Human Recombinant Erythropoietin and intravenous iron or control.

Primary end point is the amount of transfused blood. Secondary end point is the Hemoglobin level in the patient on postoperative day four.

Ancillary analysis regarding safety at 45 days and cost effectiveness are planned as well

DETAILED DESCRIPTION:
Growing evidence points out blood transfusion as a major determinant in medium and long term prognosis as regarding heart surgery population. Moreover blood has become a scarce resource, thus often delaying intervention due to lack of availability.

Previous studies at our Hospital have shown that high dose Human Recombinant Erythropoietin (HRE)effectively spares transfusions even when administered two days before surgery. The previous protocol was fragmented into 5 administration which proved to be unpractical even if effective.

After multidisciplinal discussion with nephrologists and transfusionists a new protocol was established: 80.000 UI in a single dose at time of arrival at the hospital. There are no exclusion criteria planned.

Our primary end point is the amount of transfused blood. Our secondary end point is the Hemoglobin level in the patient on postoperative day four.

Ancillary analysis regarding safety at 45 days and cost effectiveness are planned as well.

ELIGIBILITY:
Inclusion Criteria:

* All comers

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Use of allogenic blood transfusions | In hospital stay (usually 5 to 8 days after operation)

SECONDARY OUTCOMES:
Hemoglobin level on postoperative day four. | Day 4 after operation

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital, Rome, Italy

REFERENCES:
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879